CLINICAL TRIAL: NCT03777748
Title: A Pilot Study to Clinically Evaluate Maxillary and Mandibular Overdentures Retained by Two Unsplinted Diameter-reduced Titanium-zirconium Implants
Brief Title: Outcome of Implant-supported Overdentures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RWTH Aachen University (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKA 373147
Record Dates: First submitted 2018-12-06; First posted 2018-12-17 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Alveolar Bone Loss; Bone Resorption; Dental Implants; Edentulous Maxilla; Edentulous Patient
Keywords: Oral Health Impact Factor; Survival rate; Maxillary overdenture; Implant-Supported; Bone Resorption; Titanium-Zirconium; Anchor System
MeSH Terms: conditions — Alveolar Bone Loss; Bone Resorption | interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Two dental implants in the edentulous maxilla and mandible (Experimental): Edentulous maxilla und mandible are treated with two diameter-reduced tissue level implants (Straumann, Basel) and anchored with CM LOC® and CM LOC Flex® attachments (Cendres+Métaux SA, Bienne).
  Interventions: Device: dental implants and stud attachments

INTERVENTIONS:
Device: dental implants and stud attachments
  Other Names: CM LOC® and CM LOC Flex® (Cendres+Métaux SA, Bienne); (sandblasted/acid-etched) SLActive® Roxolid® implants, Ø 3.3 mm (Straumann, Switzerland)

SUMMARY:
The aim of this pilot study was to assess survival rates and peri-implant bone loss of two narrow-diameter titanium-zirconium implants supporting maxillary and mandibular overdentures during an observation time of 3 years. The masticatory performance, self-reported chewing ability and change of oral health impact profile (OHIP) after rehabilitation were also investigated.

DETAILED DESCRIPTION:
According to the recent German Oral Health Study (DMS V), toothlessness is still frequently represented in the German population. Thus in the group of 65 to 74 years old 12.4% were edentulous. Whereas in the group of 75 to 100 years old 32.8% were toothless. Toothlessness occurred more frequently in the upper jaw (19,8%) than in the lower jaw (13,7%).

Although maxillary complete dentures show less retention problems than mandibular complete dentures, edentulous patients often wish prosthesis without a palatal coverage. Since the palate is not covered by the prosthesis, the taste sense will not be affected. Zembic et al. show a significantly higher patient satisfaction for esthetics (mean difference 8.8 mm ± 24.6) and taste (mean difference 28.4 mm ± 29.9) without palatal coverage. To prevent a palatal coverage at least four implants in the upper jaw are recommended.

A systematic review concluded that implant loss rates for maxillary overdentures on two implants were significantly higher than for four implants. The recommendation to place more than two implants in the edentulous maxilla is also based on the results of a study by Richter and Knapp. Richter et al. detected very low survival rates for two implants and various anchoring elements in the edentulous upper jaw after mean observation time of five years. The 15 patients received diameter-reduced (3.25 mm) implants in the canine area. The implants were not parallel to each other due to anatomical limitations. The prostheses were attached either with telescopes or locator attachments. The implant survival rate was 39% for telescope attachments and 14% for locator attachments. The study resulted in high amount of implant fractures. In contrast, a recent study of Zembic et al. concluded an implant survival rate of 97.3% (1 year), for maxillary overdentures supported by 2 titanium-zirconium implants.

However, the systematic review and meta-Analysis from Di Francesco et al. also verifies the lack of evidence concerning the number of implants in the edentulous maxilla and the relationship between overdenture survival and the patient's quality of life.

In the planned observation study, the investigators also used diameter-reduced (3.3 mm) implants. Similarly in the study before the investigators selected a titanium-zirconium (TiZr) implant called Roxolid® (Straumann) to prevent high rate of implant fracture. According to several previous studies the TiZr small-diameter bone level implants provide at least the same outcomes after 12 month as titanium Grade IV bone level implants. The implant survival and success rates were 100% for TiZr implants.These promising results were first indications for an improved mechanical property of TiZr implants which may extend implant therapy to more challenging clinical situations, as discussed before for edentulous maxilla.

In addition, the investigators use a new anchoring system called CM LOC® and CM LOC Flex® to compensate different implant angulation. CM LOC Flex® anchor system offers the special advantage of a broad range of clinical applications due to its unique compensation function. The abutment can be angled up to 60°, which significantly reduce the wear between female part and titanium patrix. There is already an in vitro study by Passia et al., demonstrating positive long-term retention behaviour for CM LOC® in comparison to Locator anchor.

In the actual study the investigators included ten maxillary and mandible edentulous patients (58-79 years old) being dissatisfied with their complete dentures. In total, 40 diameter-reduced titanium-zirconium implants were placed in the canine region of the upper and lower jaw. Following 3 to 5 months of healing, implant-supported overdentures were inserted on two CM LOC® and CM LOC Flex® attachments depending on the indication. Implants and overdentures were evaluated at 4 weeks (baseline) and 6, 12, 24, 36 months after insertion of overdentures. Standardized radiographs were taken at implant loading and 12, 36 month after loading. Implant survival rates and bone loss were the primary outcomes.

The oral health related quality of life was assessed before and after treatment by means of the questionnaires OHIP G14. Further, each patient completed an additional questionnaire to evaluate chewing satisfaction for soft and hard foods. Questions were answered on a 100-mm visual analogue scale (VAS). Additionally, the masticatory performance was assessed with a standardized chewing test. The participants were instructed to chew standardised gums with three degrees of hardness for 30 seconds, each on the right and left side as well as on both sides. The chewed particles were then spread to a standardized detection sheet. Each sheet is placed in a tripod, and photos were made. Chewing efficacy was obtained before treatment, at baseline, 6, 12, 24, 36 month after implant loading.

Descriptive statistics were applied by calculating means, medians, standard deviations, and interquartile ranges of bone loss and of the questionnaires. Bone loss and the questionnares were statistically assessed using the Wilcoxon signed rank test. The level of significance was set at 5%.

The evaluation of the standardized masticatory function test was performed automatically through the use of a light sensor that measures the size and amounts of chewed particles.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects older than 18 years.
* Edentulous patients with a bone atrophy, which necessitates the use of diameter-reduced implants and excessive augmentation procedures are denied by the patient.
* Sufficient bone supply with minimal risk of injury to neighboring structures when using two 10 mm or longer implants per jaw.
* Bone height above the N. alveolaris inferior of at least 11 mm and the precondition of a one-stage implantation and augmentation.
* Good health condition according to the Physical Status Classification System one or two (American Society of Anesthesiologists, ASA 2010)
* Good oral hygiene and an at most moderate tobacco consumption
* Signed informed consent

Exclusion Criteria:

* Indication for large augmentations of the jaw bone
* Allergy to metallic implant components or prosthesis plastics
* Bisphosphonate therapy
* Chemo-, immuno-, or radiation therapy
* Psychological disorder
* Substance abuse
* Pregnant woman
* Persons who are placed in an institution on a judicial or administrative order
* Any other circumstances that prevent the use of oral surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Investigation of the success rates of the implants | 5 Years
  Implant fracture, implant loss
Marginal bone loss | 5 years
  Measurement of marginal bone loss on standardized radiographs [mm]

SECONDARY OUTCOMES:
Probing depth | 5 Years
  Measurement of probing depth [mm]
Gingival status | 5 Years
  Assessment of gingival index
Oral hygiene | 5 Years
  Assessment of plaque index
Oral Health Quality of Life | 5 years
  Oral Health Impact Profile - G14 (OHIP-G14, short version of the OHIP with 14 questions, according to Slade). Responses are made on a scale of never (0), hardly (1), occasionally (2), fairly often (3) and very often (4), resulting in possible values from 0 to 56 points in total.
Chewing satisfaction | 5 years
  Assessment of the chewing satisfaction using a Visual Analogue Scale (VAS). The beginning of the scale is defined as "completely dissatisfied" and the end of the line as "completely satisfied".
Masticatory performance | 5 years
  Assessment of the masticatory performance with a standardized chewing test. The participants are instructed to chew standardised gums with three degrees of hardness for 30 seconds each on the right and left sides as well as on both sides. The chewed particles were then spread to a standardized detection sheet. Each sheet is placed in a standardized stand support and are photographed.
Survival rate of prosthetic restoration | 5 years
  The prosthesis is examined for cracks, fractures, discolorations or other defects. Pass accuracy is examined. Visual and tactile control of the CM LOC® abutments and of the matrices (with retention inserts) are done.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy WM. The effect of complete dentures upon taste perception. Br Dent J. 1971 Mar 2;130(5):201-5. doi: 10.1038/sj.bdj.4802647. No abstract available. PMID 5278921
- [Background] Zembic A, Wismeijer D. Patient-reported outcomes of maxillary implant-supported overdentures compared with conventional dentures. Clin Oral Implants Res. 2014 Apr;25(4):441-50. doi: 10.1111/clr.12169. Epub 2013 Apr 15. PMID 23581398
- [Background] Roccuzzo M, Bonino F, Gaudioso L, Zwahlen M, Meijer HJ. What is the optimal number of implants for removable reconstructions? A systematic review on implant-supported overdentures. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:229-37. doi: 10.1111/j.1600-0501.2012.02544.x. PMID 23062145
- [Background] Kern JS, Kern T, Wolfart S, Heussen N. A systematic review and meta-analysis of removable and fixed implant-supported prostheses in edentulous jaws: post-loading implant loss. Clin Oral Implants Res. 2016 Feb;27(2):174-95. doi: 10.1111/clr.12531. Epub 2015 Feb 9. PMID 25664612
- [Background] Richter E, Knapp WJI. Auf zwei Eckzahnimplantaten abgestützte Oberkiefer-Coverdentureprothesen-Ergebnisse einer klinischen Studie. 2010;18:165-174.
- [Background] Zembic A, Tahmaseb A, Jung RE, Wismeijer D. One-year results of maxillary overdentures supported by 2 titanium-zirconium implants - implant survival rates and radiographic outcomes. Clin Oral Implants Res. 2017 Jul;28(7):e60-e67. doi: 10.1111/clr.12863. Epub 2016 May 6. PMID 27150942
- [Background] Al-Nawas B, Bragger U, Meijer HJ, Naert I, Persson R, Perucchi A, Quirynen M, Raghoebar GM, Reichert TE, Romeo E, Santing HJ, Schimmel M, Storelli S, ten Bruggenkate C, Vandekerckhove B, Wagner W, Wismeijer D, Muller F. A double-blind randomized controlled trial (RCT) of Titanium-13Zirconium versus Titanium Grade IV small-diameter bone level implants in edentulous mandibles--results from a 1-year observation period. Clin Implant Dent Relat Res. 2012 Dec;14(6):896-904. doi: 10.1111/j.1708-8208.2010.00324.x. Epub 2011 Mar 17. PMID 21414131
- [Background] Chiapasco M, Casentini P, Zaniboni M, Corsi E, Anello T. Titanium-zirconium alloy narrow-diameter implants (Straumann Roxolid((R))) for the rehabilitation of horizontally deficient edentulous ridges: prospective study on 18 consecutive patients. Clin Oral Implants Res. 2012 Oct;23(10):1136-41. doi: 10.1111/j.1600-0501.2011.02296.x. Epub 2011 Aug 18. PMID 22092806
- [Background] Passia N, Ghazal M, Kern M. Long-term retention behaviour of resin matrix attachment systems for overdentures. J Mech Behav Biomed Mater. 2016 Apr;57:88-94. doi: 10.1016/j.jmbbm.2015.11.038. Epub 2015 Dec 7. PMID 26705935
- [Background] Di Francesco F, De Marco G, Gironi Carnevale UA, Lanza M, Lanza A. The number of implants required to support a maxillary overdenture: a systematic review and meta-analysis. J Prosthodont Res. 2019 Jan;63(1):15-24. doi: 10.1016/j.jpor.2018.08.006. Epub 2018 Sep 28. PMID 30269880
- [Background] Jordan RA, Bodechtel C, Hertrampf K, Hoffmann T, Kocher T, Nitschke I, Schiffner U, Stark H, Zimmer S, Micheelis W; DMS V Surveillance Investigators' Group. The Fifth German Oral Health Study (Funfte Deutsche Mundgesundheitsstudie, DMS V) - rationale, design, and methods. BMC Oral Health. 2014 Dec 29;14:161. doi: 10.1186/1472-6831-14-161. PMID 25547464